CLINICAL TRIAL: NCT06542315
Title: Intraoperative Parathyroid Hormone Monitoring to Guide Surgery in Renal hyperparathyroIdism: A Pilot Trial
Brief Title: Intraoperative Parathyroid Hormone Monitoring to Guide Surgery in Renal hyperparathyroIdism
Acronym: PEREGRINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Phillip Staibano, Physician, Resident surgeon, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 151132
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Secondary Hyperparathyroidism; Tertiary Hyperparathyroidism
Keywords: hyperparathyroidism; secondary hyperparathyroidism; tertiary hyperparathyroidism; chronic kidney disease; renal transplantation; pilot trial
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Multi-arm parallel group pilot trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No IOPTH monitoring arm (No Intervention): Surgery for patients randomized to this arm will not require guidance with any IOPTH monitoring. These will be allowed to use frozen section analysis, if deemed appropriate by the surgeon.
- 10 minute arm (Experimental): Surgery for patients randomized to this arm will need to use IOPTH monitoring. Surgeons in this arm will decide to end surgery or perform surgical re-exploration if the IOPTH level at 10 minutes following ligation of all hyperfunctioning parathyroid tissue is >=50% from the highest pre-incision or pre-excision baseline IOPTH level.
  Interventions: Procedure: Intraoperative parathyroid hormone (IOPTH) monitoring
- 15 minute arm (Experimental): Surgery for patients randomized to this arm will need to use IOPTH monitoring. Surgeons in this arm will decide to end surgery or perform surgical re-exploration if the IOPTH level at 15 minutes following ligation of all hyperfunctioning parathyroid tissue is >=50% from the highest pre-incision or pre-excision baseline IOPTH level.
  Interventions: Procedure: Intraoperative parathyroid hormone (IOPTH) monitoring
- 20 minute arm (Experimental): Surgery for patients randomized to this arm will need to use IOPTH monitoring. Surgeons in this arm will decide to end surgery or perform surgical re-exploration if the IOPTH level at 20 minutes following ligation of all hyperfunctioning parathyroid tissue is >=50% from the highest pre-incision or pre-excision baseline IOPTH level.
  Interventions: Procedure: Intraoperative parathyroid hormone (IOPTH) monitoring
- 25 minute arm (Experimental): Surgery for patients randomized to this arm will need to use IOPTH monitoring. Surgeons in this arm will decide to end surgery or perform surgical re-exploration if the IOPTH level at 25 minutes following ligation of all hyperfunctioning parathyroid tissue is >=50% from the highest pre-incision or pre-excision baseline IOPTH level.
  Interventions: Procedure: Intraoperative parathyroid hormone (IOPTH) monitoring

INTERVENTIONS:
Procedure: Intraoperative parathyroid hormone (IOPTH) monitoring — Intraoperative parathyroid hormone (IOPTH) monitoring, which is a surgical adjunct that permits PTH bloodwork to be drawn during parathyroid surgery to monitor and guide surgical outcomes.
  Arms: 10 minute arm; 15 minute arm; 20 minute arm; 25 minute arm

SUMMARY:
The goal of this pilot clinical is to determine the feasibility of a fully powered clinical trial to determine the effectiveness of intraoperative parathyroid hormone (IOPTH) criteria in guiding surgery for secondary and tertiary hyperparathyroidism. The main question it aims to answer is:

Is a fully powered trial investigating the role for IOPTH criteria in secondary and tertiary hyperparathyroidism feasible?

The comparison group is surgery not guided by IOPTH.

Participants will be randomized to undergo parathyroid surgery with one of four IOPTH criteria or a control arm that does not use IOPTH. All recruited patients are asked to complete quality of life and cognitive questionnaires, in addition to bloodwork during the study period.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is increasing in prevalence globally alongside rising rates of obesity and metabolic syndromes. The rates of secondary and tertiary hyperparathyroidism are expected to rise alongside the increasing prevalence of CKD. Secondary hyperparathyroidism is diagnosed in up to 80% of patients with long-standing CKD on hemodialysis and is associated worse renal and cardiovascular outcomes and quality of life. Up to 55% of patients are non-compliant with, or refractory to, medical treatment and therefore require definitive surgery. Up to 22% of patients who undergo renal transplantation also develop tertiary hyperparathyroidism, which is associated with worse patient morbidity and renal graft outcomes. Surgery to extirpate abnormal parathyroid tissue in both diagnoses is technically challenging with surgical failure rates as high as 30%. Intraoperative parathyroid hormone (IOPTH) monitoring, which is a surgical adjunct that uses the short half-life of PTH to guide parathyroid surgery, is standard-of-care in primary hyperparathyroidism. There is no consensus nor standardization in the use of IOPTH monitoring in secondary and tertiary hyperparathyroidism. The investigators propose a multi-centre, multi-arm randomized trial to identify the most effective IOPTH monitoring criteria in improving surgical outcomes in secondary and tertiary hyperparathyroidism.

To evaluate the feasibility of a fully powered trial, the investigators will conduct a randomized and blinded multi-centre, multi-arm pilot trial. The investigators plan on evaluating five allocation arms that use four IOPTH monitoring criteria (i.e., 10 minutes, 15 minutes, 20 minutes, and 25 minutes) against a control arm of not using IOPTH monitoring. The primary feasibility outcome is randomization rate. The investigators will aim for a targeted randomization rate of 70% (95% CI: 55%-82%). Secondary feasibility outcomes include group cross-over rate, blinding effectiveness, patient compliance, and pilot trial costs. The primary efficacy outcome is recurrent hyperparathyroidism, which is evaluated at six months. Secondary efficacy outcomes will include operating room time, renal graft outcomes, renal function, cardiovascular outcomes, hospital admission and rate of re-admission, quality of life, cognitive performance. Inclusion criteria will include any adult patients (>= 18 years old) diagnosed with secondary or tertiary hyperparathyroidism who are candidates for parathyroid surgery.

The investigators plan to recruit 60 patients (12 per arm) to evaluate a randomization goal of 70% (95% CI: 55%-82%) while accounting for a 20% attrition rate. The investigators will perform descriptive analyses with ITT principles to evaluate feasibility and use these findings to evaluate the practicality of a fully powered trial. The investigators will perform descriptive analyses for all outcomes with 95% confidence intervals. The investigators will use the stop light model for determining whether a final trial is feasible, whereby a randomization rate equal to or greater than 70% will suggest that such a trial is feasible.

The results of a fully powered trial will standardize and identify the role for IOPTH monitoring in optimizing surgical outcomes for secondary and tertiary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Candidate for subtotal parathyroidectomy or total thyroidectomy with or without autotransplantation
* Tertiary hyperparathyroidism and/or recurrent hyperparathyroidism OR secondary hyperparathyroidism diagnosed with any stage of chronic kidney disease

Exclusion Criteria:

* Undergoing parathyroidectomy for primary hyperparathyroidism
* Pregnant or breastfeeding women
* Undergoing revision parathyroidectomy
* Undergoing minimally invasive or video-assisted parathyroidectomy
* Unable to provide written consent to be participant in study
* Unable to complete study follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Randomization rate | From enrollment to the end the trial at 6 months
  Defined as the number of patients agreeing to participate in the trial and being randomized to any of the allocation groups, divided by the number of eligible patients. We will review this data every two weeks during the pilot trial. A randomization percentage of 70% or greater will support the feasibility of a fully powered RCT. We will utilize the traffic light system introduced by Avery and colleagues, whereby if randomization of 70% or greater is achieved, we will proceed with fully powered trial. If a randomization rate of 50-69% is achieved, we will consider proceeding with modifications to the fully powered trial. If randomization rate is <50%, we will not proceed with fully powered trial. We selected this as a primary feasibility outcome because we are sampling from a relatively rare population, and so gathering an accurate estimate of randomization rate will allow us to determine the ideal number of participating sites for the final trial.

SECONDARY OUTCOMES:
Blinding effectiveness | From enrollment to the end the trial at 6 months
  The Bang Blindness Inventory (BBI) will be administered to patients, outcome assessors, and statisticians at the end of study follow-up and the time of trial completion (for statisticians). The BBI will then be calculated for each of these blinded parties and reported on a scale of -1 (unblinding) to 0 (perfect blinding) to +1 (lack of blinding).
Surgeon compliance and crossover | From enrollment to the end the trial at 6 months
  Surgeon compliance and crossover: The number of patients who undergo surgery with a different IOPTH monitoring criteria from which they were randomized. All surgeons will complete a postoperative de-brief form that will capture their rationale for changing groups. We will consider any percentage of group crossover to hinder consideration of a fully powered trial and based on the direction and number of groups crossovers. If any crossovers are detected, then we will consider to the number and organization of allocation arms for the fully powered trial.
Follow-up completion | From enrollment to the end the trial at 6 months
  Defined as completion of all questionnaires and study bloodwork from randomization to final study follow-up.
Trial costs | From enrollment to the end the trial at 6 months
  We will estimate the study and hospital costs required for this multi-centre initiative for each recruited patient during the study period. This will provide an estimate of the costs for performing the fully powered trial.

OTHER OUTCOMES:
Surgeon-dictated changes to intraoperative plan | From enrollment to the end the trial at 6 months
  Any changes to the surgical plan will be documented by surgeons in a postoperative de-brief form.
Operating time | From enrollment to the end the trial at 6 months
  The length of the surgery from skin incision to skin closure, as measured in minutes
Revision surgery rate and indication for revision surgery | From enrollment to the end the trial at 6 months
  Number of patients who either undergo or are consented and scheduled to undergo revision parathyroidectomy within 6 months of randomization. This will be measured as a dichotomous outcome. We will also evaluate the surgical indication for revision surgery. This will be measured as a categorical outcome.
Chronic kidney disease progression, cardiovascular death, or renal death (composite outcome) | From enrollment to the end the trial at 6 months
  Number of patients who meet the criteria of this composite outcome (sustained decline in eGFR of at least 50%, end-stage kidney disease, or kidney-related or cardiovascular death).
Recurrent and/or persistent hyperparathyroidism rates | From enrollment to the end the trial at 6 months
  Number of people who continue to have pathologically elevated PTH levels within 3 months of randomization. This will be measured with reference to the defined PTH reference threshold at each participating institution. This will be measured immediately after surgery and at one month and six months from randomization. We will also measure the number of patients who have laboratory hypercalcemia as defined by bloodwork immediately after surgery and at one month and six months from randomization.
IOPTH kinetics in secondary and tertiary hyperparathyroidism | From enrollment to the end the trial at 6 months
  The IOPTH change (as a percent) between time points will be described.
Emergency room visits and hospital readmission rates | From enrollment to the end the trial at 6 months
  Number of emergency room visits and hospital readmissions due to surgical complications.
Length of hospital stay | From enrollment to the end the trial at 6 months
  Number of days admitted to hospital from the date of surgery to the day of hospital discharge. We will also measure the length of hospital stay for any readmissions from hospital admission to discharge.
Health-related quality of life | From enrollment to 3 months
  These will be measured using the SF-36 tool and kidney disease quality of life (KDQOL)-36 tool prior to randomization (baseline), and at one month and three months from surgery. The SF-36 is a validated self-reported patient-centred outcome measure (PROM) measured via eight domains on a 0-100 scale with lower scores indicating worse disability. The KDQOL-36 is a validated self-reported PROM scored from 0-100 with higher scores indicating better quality of life.
Renal graft failure and renal graft complication rates | From enrollment to the end the trial at 6 months
  Number of patients who have renal transplantation who experienced renal graft failure and/or complication during the study period.
Rates of hypoparathyroidism and hypocalcemia | From enrollment to the end the trial at 6 months
  These will be measured by calculating the number of patients who develop hypoparathyroidism and/or hypocalcemia following surgery.
Surgery-specific complication rates | From enrollment to the end the trial at 6 months
  The types of surgical complications will be documented.
Fully powered trial costs | From enrollment to the end the trial at 6 months
  This will be collected during the study period. It will include operative and inpatient/outpatient costs for each randomized patient.
Cognitive function | From enrollment to 3 months
  These will be measured using the Hospital Anxiety and Depression Scale (HADS) and MoCA prior to randomization (baseline), and at one month and three months postoperatively. In the HADS, higher scores indicate worse anxiety and depression scores with scores ranging from 0-21. In the MoCA, lower scores indicate worse cognitive function with scores ranging from 0-30.

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This will need to be further discussed with all trial team members prior to making final decision.

REFERENCES:
- [Result] Kovesdy CP. Epidemiology of chronic kidney disease: an update 2022. Kidney Int Suppl (2011). 2022 Apr;12(1):7-11. doi: 10.1016/j.kisu.2021.11.003. Epub 2022 Mar 18. PMID 35529086
- [Derived] Staibano P, Au M, Pasternak JD, Parpia S, Zhang H, Busse JW, Nguyen NT, Monteiro E, Gupta MK, Choi DL, Lewis T, McKechnie T, Thabane A, Ham J, Young JE, Bhandari M. Intraoperative parathyroid hormone monitoring to guide surgery in renal hyperparathyroidism (PEREGRINE): a protocol for a randomised multiarm surgical pilot trial. BMJ Open. 2025 Jul 17;15(7):e098860. doi: 10.1136/bmjopen-2025-098860. PMID 40675640